CLINICAL TRIAL: NCT04902053
Title: INSPIRIS RESILIA Aortic Valve, Valve-in-Valve Surveillance Study
Acronym: INVIVITY
Status: Suspended | Type: Observational
Why Stopped: Lack of enrollment. Study will be restarted when there is sufficient INSPIRIS Valve in Valve case volume to support enrollment.
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-12
Record Dates: First submitted 2021-05-12; First posted 2021-05-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Aortic Valve Replacement
Keywords: INVIVITY; RESILIA; INSPIRIS; Valve in Valve; TAVR; Aortic Transcatheter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Subjects previously implanted with INSPIRIS RESILIA Model 11500A and are undergoing planned valve-in-valve treatment. — Designed to capture Adverse Event information and valve measurement data from dysfunctional INSPIRIS RESILIA aortic valves before and after Valve-in-valve (ViV) treatment.

SUMMARY:
The primary objective of the INSPIRIS RESILIA Aortic Valve-in-valve (ViV) Surveillance Study ("the Study") is to capture Adverse Event information and valve measurement data from dysfunctional INSPIRIS RESILIA aortic valves before and after Valve-in-valve (ViV) treatment.

DETAILED DESCRIPTION:
This is a single-arm observational study which includes both prospective and retrospective data.

At least fifty (50) Subjects enrolled prospectively prior to the ViV procedure, or retrospectively after the ViV procedure (within 37 days post-ViV procedure) with dysfunctional 19mm-25mm INSPIRIS aortic valves, will participate in this study.

All subjects will be followed for up to 1 month after the TAVR ViV procedure.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following Inclusion Criteria:

1. 18 years or older at the time of the TAVR ViV treatment
2. Has an INSPIRIS RESILIA aortic valve implanted in the aortic position confirmed to be size 19mm, 21mm, 23mm or 25mm
3. A ViV procedure using an Edwards transcatheter aortic heart valve (TAVR) has been scheduled; or completed within 37 days from time of consent
4. The participant agrees to attend a follow-up assessment at 1 month post ViV procedure
5. The participant provides written informed consent prior to the post-ViV procedure CT scan

Exclusion Criteria:

Subjects must not meet any of the following Exclusion Criteria:

1. The INSPIRIS RESILIA aortic valve size is

   * Unconfirmed, or
   * Confirmed to be 27mm or 29mm
2. Prior re-interventions have been performed on the INSPIRIS RESILIA aortic valve
3. The INSPIRIS RESILIA aortic valve has been subjected to balloon aortic valvuloplasty (BAV) prior to the baseline quantitative area measurement of the valve area
4. The Subject is pregnant or desires to become pregnant within 40 days of the ViV procedure
5. Subjects with a known contraindication or hypersensitivity to contrast media that cannot be adequately pre-medicated per hospital guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously implanted with INSPIRIS RESILIA Model 11500A and are undergoing planned valve-in-valve treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2028-06 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Subject's Occurrence Rate of the Composite Safety Endpoint | Events occurring within 30 days of valve-in-valve procedure
  The primary safety endpoint is a composite endpoint defined as all-cause mortality, all stroke (disabling and non-disabling), life-threatening bleeding, new requirement for dialysis, coronary artery compression or obstruction, major vascular complication, and valve-related dysfunction requiring reintervention.
  Data will be reported as the number (and percent) of subjects who experience an event divided by the number of enrolled subjects times 100.
Subject's Occurrence Rate of Valve Malpositioning | Events occurring within 30 days of valve-in-valve procedure
  Valve malpositioning includes all instances of ViV-TAVR migration, embolization, and valve recapture or retrieval.
  Data will be reported as the number (and percent) of subjects who experience an event divided by the number of enrolled subjects times 100.
Subject's INSPIRIS RESILIA Valve Expansion Post Valve in Valve Procedure Compared to Baseline | Day 30, compared to baseline
  A primary effectiveness endpoint is the expansion, measured in mm^2, of INSPIRIS valve for sizes 19mm-25mm, following the Edwards transcatheter aortic valve implantation.

SECONDARY OUTCOMES:
Subject's Occurrence Rate of Reportable Adverse Events | Events occurring within 30 days of valve-in-valve procedure
  Reportable Adverse Events mirroring those being reported to the STS/ACC TVT Registry.
  Data will be reported as the number (and percent) of subjects who experience an event divided by the number of enrolled subjects times 100.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Johnston, MD, FACS, Principal Investigator — Northwestern University
Locations (7):
- United States (7):
  - University of Southern California, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - St. Vincent Hospital, Indianapolis, Indiana
  - Nyph/Cumc, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.